CLINICAL TRIAL: NCT03681301
Title: Development and Impact Assessment of Virtual Reality Simulator on the Education of the Endotracheal Intubation in the Medical Students
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Early Terminated
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 4-2018-0571
Record Dates: First submitted 2018-09-20; First posted 2018-09-24 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Medical Education
MeSH Terms: interventions — Intubation, Intratracheal

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Investigator, Outcomes Assessor
Masking Description: Double (Investigator, Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional (Experimental): Additional self-directed learning and practice using virtual reality simulator, after conventional training session
  Interventions: Other: virtual reality simulator
- Control (No Intervention): Conventional training session which includes didactic teaching and low-fidelity simulation session involving trainer's demonstration, followed by hands-on practice

INTERVENTIONS:
Other: virtual reality simulator — Additional self-directed learning and practice using virtual reality simulator
  Other Names: virtual reality simulator for endotracheal intubation
  Arms: Interventional

SUMMARY:
The medical school educates students on essential skills, which is an important task. Especially, endotracheal intubation is considered an important option in the management of cardiopulmonary resuscitation.

To avoid technical and ethical concerns of training involving real patients, conventional teaching methods incorporate the use of a low-fidelity manikin in replacement. However, the manikin anatomy often lacks the realism of a live human.

The addition of virtual reality technology may optimize learning by providing an ethical, cost-effective and more realistic modality to acquire the basic skills of intubation. If it is proven to be effective, efforts to integrate virtual reality technology into routine training of such procedures in the medical school should be promoted.

The investigators hypothesize that the addition of virtual reality mobile application to conventional training will improve procedural skill dexterity and proficiency and hence, improve learner's satisfaction and confidence in performing endotracheal intubation.

ELIGIBILITY:
Participants included medical school students without intubation intubation experience

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2019-08-03 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Total score of required 20-key points of intubation during endotracheal intubation procedure | within 1 month after training session
  During the intubation training evaluation using manikin, the score was added by using the check list Which is consisted of the patient's positioning, opening the mouth, laryngoscope handling, glottis view evaluation, insertion and fixation of the endotracheal tube, etc, and consists of a total of 20 points

SECONDARY OUTCOMES:
Intubation complete time (secs) | within 1 months after training session
  Impact assessment of virtual reality simulator for endotracheal intubation
Overall proficiency grading (fail/ pass/ high pass/ honors) | within 1 months after training session
  Impact assessment of virtual reality simulator for endotracheal intubation
Overall confidence, anxiety, comfort level: 5-point Likert scale (1 = very low, 2 = low, 3 = moderate, 4 = high, 5 = very high) | within 1 months after training session
  Impact assessment of virtual reality simulator for endotracheal intubation

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Anesthesia and Pain Research Institute, Yonsei University College of Medicine, Seoul, South Korea